CLINICAL TRIAL: NCT05100043
Title: IL-4 and IFN-γ As Immunologic Predictors of Response to HPV Immunotherapy in Warts
Brief Title: Interleukin 4 and Interferon Gamma Predictors of Human Papillomavirus Immunotherapy in Warts
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Noha M Hammad, MD, Principal investigator, Zagazig University
Other Study IDs: 3140-23-10-2019
Record Dates: First submitted 2021-10-05; First posted 2021-10-29 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Warts Hand; Wart, Genital
MeSH Terms: conditions — Condylomata Acuminata | interventions — Interleukin-4

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cases: Patients having multiple recurrent and recalcitrant cutaneous and genital warts
  Interventions: Biological: IL-4 and IFN-γ measurements
- Controls: Healthy volunteers matched for age and sex
  Interventions: Biological: IL-4 and IFN-γ measurements

INTERVENTIONS:
Biological: IL-4 and IFN-γ measurements — Blood samples are withdrawn from participants and whole blood cultures are prepared and stimulated by bivalent HPV vaccine.IL-4 and IFN-γ are measured in culture supernatants

SUMMARY:
In the present study the investigators assessed the invitro role of IL-4 and IFN-γ in predicting the response to bivalent HPV vaccine after whole blood stimulation

DETAILED DESCRIPTION:
40 Patients and 40 controls are enrolled in the study. Participants suffer from chronic recurrent cutaneous and genital warts. Blood samples were withdrawn then whole blood cultures are prepared. Cultures are stimulated with bivalent HPVvaccine. IL-4 and IFN-γ measurement in culture supernatants by ELISA. IL-4 and IFN-γ are investigated to predict the therapeutic response to bivalent HPV vaccine immunotherapy in warts.

ELIGIBILITY:
Inclusion Criteria:

* Patients with recurrent and recalcitrant cutaneous and anogenital warts.

Exclusion Criteria:

* History of allergy to the HPV vaccine
* Active viral, fungal, or bacterial infections
* Immunosuppressive diseases or drugs.
* Autoimmune diseases, or other systemic diseases, e.g., hepatic, or renal disorders, diabetes, meningitis or convulsions
* Skin allergies
* Pregnancy and lactation
* Earlier wart treatment at least one month before enrollment.

Min Age: 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients are attendants in Zagazig University Hospitals Dermatology outpatient clinic
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-01-03 (Actual); Primary Completion 2020-07-03 (Actual); Study Completion 2021-03-02 (Actual)

PRIMARY OUTCOMES:
Change of IFN-γ and IL-4 levels | 48 hours
  Quantitative measurement of IFN-γ and IL-4 in culture supernatants

SECONDARY OUTCOMES:
Change in the size of warts | 6 months
  Clinical observation and photographing of wart size

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Marei, MD, PhD, Study Director — Faculty of Medicine, Zagazig University , Zagazig, Egypt
Locations (1):
- Zagazig University Faculty of Medicine, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: Undecided